CLINICAL TRIAL: NCT06434870
Title: Comparison of the Effect of Spinal Anesthesia Applied in Elective Cesarean Cases on Frontal QRS Angle in Anemic and Non-Anemic Patients
Brief Title: Effect of Spinal Anesthesia in Elective Cesarean Cases on Frontal QRS Angle in Anemic and Non-Anemic Patients
Status: Recruiting | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, ahmet kaya, assistant professor, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: MAIEAH630004
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Anemia; Electrocardiography; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who had undergone Elective Cesarean Surgery with anemia: In pregnant women, haemoglobin values below 11 mg/dL in the first trimester, 11 mg/dL in the second trimester and 10.5 mg/dL in the third trimester indicate anaemia.
  The group comprised patients with haemoglobin levels below 10.5 mg/dL.
- Patients who had undergone Elective Cesarean Surgery without anemia: In pregnant women, haemoglobin values below 11 mg/dL in the first trimester, 11 mg/dL in the second trimester and 10.5 mg/dL in the third trimester indicate anaemia.
  The group comprised patients with haemoglobin levels above 10.5 mg/dL.

SUMMARY:
The QRS-T angle represents a novel marker of myocardial repolarisation. It is defined as the angle difference between the direction of ventricular depolarisation (QRS wave) and the direction of ventricular repolarisation (T wave). It is an indicator of instability in the electrophysiological properties of the myocardium and is associated with arrhythmias. The frontal QRS-T angle is a straightforward, cost-effective parameter that can be readily obtained from 12-lead electrocardiography.

The most prevalent arrhythmias during pregnancy are atrial arrhythmias. However, ventricular tachyarrhythmias are exceedingly rare during pregnancy and may be life-threatening.

Caesarean section is one of the most common surgical procedures. General anaesthesia, spinal anaesthesia and epidural anaesthesia can be employed in these patients. Spinal anaesthesia is a frequently employed method in caesarean section operations due to its rapid onset of effect, technical simplicity of application and higher probability of success.

In pregnant women, anaemia is defined as a haemoglobin concentration below 11 mg/dL in the first trimester, 11 mg/dL in the second trimester and 10.5 mg/dL in the third trimester.

DETAILED DESCRIPTION:
The QRS-T angle represents a novel marker of myocardial repolarisation. It is defined as the angle difference between the direction of ventricular depolarisation (QRS wave) and the direction of ventricular repolarisation (T wave). It is an indicator of instability in the electrophysiological properties of the myocardium and is associated with arrhythmias. The frontal QRS-T angle is a straightforward, cost-effective parameter that can be readily derived from 12-lead electrocardiography. The angle between the QRS and T waves is a useful indicator of myocardial repolarisation. It is associated with arrhythmias and instability in the electrophysiological properties of the myocardium. The frontal QRS-T angle is a simple, inexpensive parameter that can be easily obtained from 12-lead electrocardiography.

Pregnancy has a profound effect on the cardiovascular system. It results in an increase in blood volume, heart rate, venous pressure in the lower extremities, and cardiac output. Furthermore, it can result in a reduction in peripheral resistance and pulmonary vascular resistance, as well as a decline in blood pressure. Furthermore, it affects the cardiac conduction system, rendering patients more susceptible to arrhythmias. The most prevalent arrhythmias during pregnancy are atrial arrhythmias. Ventricular tachyarrhythmias are relatively uncommon during pregnancy and can be life-threatening.

One of the most common surgical procedures is caesarean section. General anaesthesia, spinal anaesthesia and epidural anaesthesia can be employed in these patients. Spinal anaesthesia is a frequently employed method in caesarean section operations due to its rapid onset of effect, technical ease of application and higher chance of success. In addition to the beneficial effects, direct cardiac and indirect cardiac side effects may be observed, such as vasodilatation due to sympathetic denervation, decreased right heart pressure and reflex bradycardia, which depend on the level of block.

In pregnant women, haemoglobin values below 11 mg/dL in the first trimester, 11 mg/dL in the second trimester and 10.5 mg/dL in the third trimester are considered to indicate anaemia.

The objective of this study was to investigate the effects of spinal anaesthesia in elective caesarean section cases on frontal QRS angle in anaemic and non-anaemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Patients with American Society of Anesthesiologists (ASA) II classification

Exclusion Criteria:

* Patients with rhythm disorders
* Patients with electrolyte disturbances
* Patients with liver and/or renal failure
* Obese patients (body mass index > 30)
* Trauma patients
* Cancer patients
* ASA III-IV patients
* Patients who do not wish to participate in the study will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include 100 patients aged 18-45 years with an American Society of Anesthesiologists (ASA) II classification who will undergo elective caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The measurements to be taken include QRS, frontal QRS, QRS angle and Tp-e interval. (T1) | preoperatively
The measurements to be taken include QRS, frontal QRS, QRS angle and Tp-e interval.(T2) | after spinal anaesthesia
The measurements to be taken include QRS, frontal QRS, QRS angle and Tp-e interval.(T3) | 5 min after spinal anaesthesia
The measurements to be taken include QRS, frontal QRS, QRS angle and Tp-e interval.(T4) | 5 min after spinal anaesthesia
The measurements to be taken include QRS, frontal QRS, QRS angle and Tp-e interval.(T5) | 10 min after spinal anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Turkey Sanliurfa Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)